CLINICAL TRIAL: NCT03308188
Title: EMPOWER: Evaluating the Ability to Reduce Morphine Equivalent Dose for Chronic Pain Patients Receiving Opioid-therapy Through a Web-based E-Health Self-management Program: a Randomized Multi-site Clinical Trial in Primary Care
Brief Title: EMPOWER: Randomized Trial of Online Chronic Pain Management Program to Reduce Reliance on Opioid Analgesic Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, T. John Winhusen, PhD, Professor; Vice Chair and Division Director of Addiction Sciences, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-2301; 1R01DA044248-01 (NIH)
Record Dates: First submitted 2017-10-06; First posted 2017-10-12 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Pain
Keywords: Opioid therapy; web-based intervention; self-management
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (No Intervention): Participants randomized to Treatment As Usual will receive treatment for chronic pain as typically provided by their clinician -- they will receive no extra treatment from the study.
- E-Health+ (Experimental): Participants randomized to the E-health+ arm will receive treatment as typically provided by their clinician plus a 4-month subscription to the E-health program, which is an internet based chronic pain program.
  Interventions: Behavioral: E-health program

INTERVENTIONS:
Behavioral: E-health program — The Goalistics Chronic Pain Management Program, referred to as the E-health program in EMPOWER, was developed from cognitive, behavioral, interpersonal, and self-management interventions with demonstrated efficacy in traditional face-to-face or group settings. It is patient-centered, having been developed based on substantial input from people with chronic pain and chronic pain professionals.
  Arms: E-Health+

SUMMARY:
This is a 10-month internet-based randomized controlled trial to evaluate whether an online chronic pain management program ("E-Health") can assist with reduced opioid reliance in chronic pain patients. About half of the eligible participants will receive access to the E-Health program in addition to their standard chronic pain treatment; the other half will just continue receiving their standard chronic pain treatment.

DETAILED DESCRIPTION:
This study will determine whether an innovative, accessible E-health intervention can assist with reduced opioid reliance in chronic pain patients, which can, ultimately, reduce risks of unintended opioid overdose and death. Importantly, the study will contribute to a better understanding of the mechanisms contributing to opioid use reduction while managing pain. The findings may assist in developing treatment options for a population at risk for opioid adverse effects.

Potential participants will be identified through electronic health record (EHR) queries at participating sites. Participants will be assessed at baseline, at the end of the 4-month treatment period, and at 6 months following end-of-treatment through an electronic data capture system accessed by the participants. Other outcome data will be obtained from the participant's EHR data.

ELIGIBILITY:
Inclusion Criteria:

* Be 25-80 years of age
* Be able to understand the study, and having understood, provide informed consent in English
* Have a daily average prescribed MED ≥ 20 mg over a recent three-month period
* Have a chronic pain-related diagnosis
* Self-report current use of opioid medication(s) to treat pain
* Have a Brief Pain Inventory Pain Intensity score ≥3
* Have internet access and a working email account

Exclusion Criteria:

* Be anyone who, in the judgment of study staff, would be unlikely to complete the study (e.g., planning to change to a different primary care clinic, have a terminal illness, etc.)
* Be unwilling/unable to complete the WebNeuro assessments
* Be pregnant
* Be a prisoner

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, Ph.D., Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - Duke Health, Durham, North Carolina
  - UC Health, Cincinnati, Ohio

REFERENCES:
- [Derived] Wilson M, Dolor RJ, Lewis D, Regan SL, Vonder Meulen MB, Winhusen TJ. Opioid dose and pain effects of an online pain self-management program to augment usual care in adults with chronic pain: a multisite randomized clinical trial. Pain. 2023 Apr 1;164(4):877-885. doi: 10.1097/j.pain.0000000000002785. Epub 2022 Sep 15. PMID 36525381

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment As Usual | E-Health+
Started | 202 | 200
Completed | 202 (The baseline morphine equivalent dose for one participant was an unusable outlier. MED, morphine equivalent dose; TAU, treatment as usual.) | 196
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment As Usual | E-Health+ | Total
Number analyzed (Participants) | 202 | 200 | 402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 155 | 160 | 315
  >=65 years | 47 | 40 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (10.9) | 56.4 (11.1) | 56.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 139 | 279
  Male | 62 | 61 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 189 | 191 | 380
  Unknown or Not Reported | 11 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 29 | 43 | 72
  White | 154 | 147 | 301
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 11 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 202 | 200 | 401
Morphine Equivalent Dose (MED) [Mean (Standard Deviation); unit: Morphine Equivalent Dose] — Population: Measure Analysis Population Description: The baseline morphine equivalent dose for one participant was an unusable outlier. MED, morphine equivalent dose (Treatment as Usual)
  Morphine Equivalent Dose
    number analyzed (Participants) | 201 | 200 | 401
    (all) | 47.8 (53.4) | 48.1 (63.6) | 48.0 (58.6)
Pain Intensity [Mean (Standard Deviation); unit: Score on a scale] — The Brief Pain Inventory, Pain Intensity Subscale, range: 0-10, higher values indicate more intense pain, Mean (SD)
  Score on a scale | 5.9 (1.6) | 5.9 (1.5) | 5.9 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Morphine Equivalent Dose (MED)
Description: Whether (yes/no) there was a ≥15% decrease in MED, between baseline and 10-month post-randomization follow-up.
Time Frame: Baseline and 10 months
Population: Three participants withdrew consent. (E-Health) One participant died. (E-Health) The baseline morphine equivalent dose for one participant was an unusable outlier. MED, morphine equivalent dose (Treatment as Usual)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual | E-Health+
Number analyzed (Participants) | 201 | 196
Participants | 85 | 105

2. Secondary Outcome: Pain Intensity
Description: Whether (yes/no) there is a clinically meaningful decrease in pain intensity (at least 2 points) as measured by the Brief Pain Inventory (BPI), between baseline and 10-month post-randomization follow-up.
Time Frame: Baseline and 10 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment As Usual | E-Health+
Number analyzed (Participants) | 201 | 196
Participants | 13 | 24

ADVERSE EVENTS:
Time Frame: Randomization through Month 10
Description: A potential AE is defined as >30% symptom deterioration from baseline as indicated by any of the following: 1) Pain Intensity score or Pain Interference score as measured by the BPI; 2) Depression, Anxiety, or Stress score from the DASS-21. Additionally, to meet criteria for an AE, these follow-up scores must fall within at least the "moderate" range of severity for the respective measures. A report identifying participants with AEs defined as above was generated on a weekly basis.
Arm/Group | Treatment As Usual | E-Health+
All-Cause Mortality (participants affected / at risk) | 0/202 | 1/200
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/200
Other Adverse Events (participants affected / at risk) | 95/202 | 85/200
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment As Usual (N=202) | E-Health+ (N=200)
Worsening of Pain Intensity (General disorders) | 21 | 18 — Per BPI
Worsening of Pain Interference (General disorders) | 35 | 29 — Per BPI
Worsening of Depression (Psychiatric disorders) | 37 | 30 — Per DASS-21
Worsening of Anxiety (Psychiatric disorders) | 36 | 39 — Per DASS-21
Worsening of Stress (Psychiatric disorders) | 20 | 23 — Per DASS-21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03308188/Prot_SAP_000.pdf